CLINICAL TRIAL: NCT05573035
Title: A Phase 1 Study to Assess the Safety and Efficacy of LYL845 in Adults With Relapsed and/or Refractory Metastatic or Locally Advanced Melanoma and Selected Solid Tumor Malignancies
Brief Title: A Study to Investigate LYL845 in Adults With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pipeline Reprioritization
Sponsor: Lyell Immunopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYL845-101
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Melanoma; Non-small Cell Lung Cancer; Colorectal Cancer
Keywords: TIL; tumor infiltrating lymphocyte; melanoma; non-small cell lung cancer; colorectal cancer; NSCLC; CRC; relapsed; refractory; locally advanced; advanced; metastatic; epigenetic
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label, dose-escalation and -expansion study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental LYL845 (Experimental): Epigenetically reprogrammed tumor infiltrating lymphocyte (TIL) therapy
  Interventions: Biological: LYL845

INTERVENTIONS:
Biological: LYL845 — LYL845 is an autologous tumor infiltrating lymphocyte (TIL) enhanced via Epi-R, a proprietary epigenetic reprogramming technology

SUMMARY:
This is an open-label, multi-center, dose-escalation study with expansion cohorts, designed to evaluate the safety and anti-tumor activity of LYL845, an epigenetically reprogrammed tumor infiltrating lymphocyte (TIL) therapy, in participants with relapsed or refractory (R/R) metastatic or locally advanced melanoma, non-small cell lung cancer (NSCLC), and colorectal cancer (CRC).

DETAILED DESCRIPTION:
This is an open-label, multi-center, dose-escalation study with expansion cohorts, designed to evaluate the safety and anti-tumor activity of LYL845, an epigenetically reprogrammed tumor infiltrating lymphocyte (TIL) therapy, in participants with relapsed or refractory (R/R) metastatic or locally advanced melanoma, non-small cell lung cancer (NSCLC), and colorectal cancer (CRC). During the dose-escalation phase of the study (Part A), participants with melanoma will be enrolled. Once a safe recommended Phase 2 dose range (RP2DR) has been established in Part A, enrollment will be expanded (Part B) to include additional participants with melanoma, NSCLC and CRC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years up to ≤ 75 years at the time of informed consent
* Confirmed diagnosis of melanoma, non-small cell lung cancer (NSCLC), or colorectal cancer (CRC) that is metastatic or locally advanced or unresectable and is relapsed and/or refractory (R/R) after standard therapy for each tumor histology
* Participants must have received prior systemic treatment for their metastatic disease or locally advanced disease based on tumor type as follows:
* Melanoma: participants with disease progression following an immune checkpoint inhibitor (CPI)
* NSCLC: participants with disease progression following at least 1 approved systemic therapy, including an immune CPI-containing regimen for appropriate patients or an approved targeted therapy for known molecular abnormalities if applicable to their disease
* CRC: participants with disease progression following at least 1 line of therapy, including a fluoropyrimidine with oxaliplatin or irinotecan. Microsatellite instability (MSI) high/mismatch repair deficient (dMMR) CRC participants must have disease progression following systemic therapy with immune CPIs.
* Measurable disease including at least 1 lesion that is safely resectable AND a target lesion to measure response and an additional lesion for biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ and marrow function
* Women of childbearing potential must have a negative pregnancy test at screening
* All participants must agree to practice highly effective methods of contraception
* Fully recovered from toxicity from prior systemic anticancer therapy

Exclusion Criteria:

* Prior treatment with adoptive cellular therapy
* Prior solid organ transplantation
* Central nervous system (CNS) involvement of disease that is extensive, symptomatic or untreated, or patients with leptomeningeal disease
* Uncontrolled or symptomatic pleural effusion or ascites
* Untreated or active systemic infection
* Active autoimmune disease requiring treatment or primary immunodeficiency syndrome
* Systemic corticosteroids at a dose of >10 mg of prednisone or equivalent per day
* Other primary malignancy within 3 years prior to enrollment
* Impaired cardiac function or clinically significant cardiovascular disease
* Required chronic anticoagulation, such as warfarin, low molecular weight heparin, or Factor Xa inhibitors
* Pregnant or nursing (lactating) women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Up to 28 days
  Evaluate incidence of dose-limiting toxicities (DLTs)
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years
  Evaluate incidence of treatment-emergent adverse events (TEAEs)
Severity of treatment-emergent adverse events (TEAEs) | Up to 2 years
  Evaluate severity of treatment-emergent adverse events (TEAEs)
Determine recommended Phase 2 Dose Range (RP2DR) | Up to 2 years
  Determine the recommended Phase 2 dose range (during dose-escalation phase)

SECONDARY OUTCOMES:
Overall response rate (ORR) by RECIST, version 1.1 | up to 2 years
  Evaluate anti-tumor activity of LYL845 based on overall response rate (ORR) by RECIST, version 1.1
Duration of response (DOR) | up to 2 years
  Evaluate duration of response (DOR)
Progression-free survival (PFS) | up to 2 years
  Evaluate progression-free survival (PFS)
Overall survival (OS) | up to 2 years
  Evaluate overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - UC Davis Coomprehensive Cancer Center, Sacramento, California
  - UCLA Medical Center, Santa Monica, California
  - Stanford University, Stanford, California
  - Yale Cancer Center, Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Comprehensive Cancer Center, Rochester, Minnesota
  - Hackensack Meridian Health Inc, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No